CLINICAL TRIAL: NCT06911320
Title: A Phase 1, Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Safety and Pharmacokinetics of Bemnifosbuvir and Ruzasvir Administered as a Fixed-Dose Combination in Adult Participants With Severe Renal or Hepatic Impairment in Comparison to Healthy Participants
Brief Title: Study of Bemnifosbuvir/Ruzasvir as a Fixed-dose Combination in Subjects With Normal or Severely Impaired Renal or Hepatic Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-010
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteer Study; Hepatic Impairment; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — AT-511

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 - Severe Renal Impairment (Experimental): Single dose Bemnifosbuvir (BEM)/Ruzasvir (RZR) as a fixed-dose combination
  Interventions: Drug: Bemnifosbuvir (BEM)/Ruzasvir (RZR) as a fixed-dose combination
- Group 2 - Severe Hepatic Impairment (Experimental): Single dose Bemnifosbuvir (BEM)/Ruzasvir (RZR) as a fixed-dose combination
  Interventions: Drug: Bemnifosbuvir (BEM)/Ruzasvir (RZR) as a fixed-dose combination
- Group 3 - Matched Healthy Subjects (Experimental): Single dose Bemnifosbuvir (BEM)/Ruzasvir (RZR) as a fixed-dose combination
  Interventions: Drug: Bemnifosbuvir (BEM)/Ruzasvir (RZR) as a fixed-dose combination

INTERVENTIONS:
Drug: Bemnifosbuvir (BEM)/Ruzasvir (RZR) as a fixed-dose combination — A single dose of BEM/RZR will be administered
  Other Names: AT-527 (BEM) and AT-038 (RZR)

SUMMARY:
To Assess the Effect of Severe Hepatic or Renal Impairment on the Pharmacokinetics of Bemnifosbuvir/Ruzasvir After a Single Dose

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* BMI of 18.5 to 43.0 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Renal Impaired Subjects (Group 1):

* Considered stable in the judgement of an Investigator
* Presence of severe renal impairment or kidney failure (as defined by eGFR< 30 mL/ min)

Hepatic Impaired Subjects (Group 2):

* Considered stable for at least 1 month prior to Screening, as per the judgement of an Investigator
* Presence of severe hepatic impairment (Child-Pugh Class C: score of 10 to 15).

Subjects with Normal Hepatic and Renal Function (Group 3):

* Medically healthy, in the opinion of an Investigator
* Must match by gender, age (± 10 years), and BMI (within 20%) to the pooled mean values of subjects with severe renal and hepatic impairment

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with hepatitis B virus, hepatitis C virus or HIV
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Renal and Hepatic Impaired Subjects (Group 1 and 2):

* Presence of poorly controlled Type 1 or Type 2 diabetes as defined by Hemoglobin A1c > 10%
* Undergoing any method of dialysis
* Subjects requiring treatment for hepatic impairment or other chronic disease must be on a stable treatment plan

Renal Impaired Subjects (Group 1):

* History of renal transplant
* Concurrent use of medications known to affect the elimination of serum creatinine

Hepatic Impaired Subjects (Group 2):

* History of liver transplant
* Evidence of hepatic carcinoma presence at Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of BEM/RZR Maximum plasma concentration (Cmax) | Day 1
Pharmacokinetics (PK) of BEM/RZR Area under the plasma concentration-time curve (AUC) | Day 1
Pharmacokinetics (PK) of BEM/RZR AUC | Day 1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atea Study Site, Orlando, Florida
  - Atea Study Site, Tampa, Florida